CLINICAL TRIAL: NCT00594750
Title: Mechanisms of Exacerbation of Asthma
Acronym: MECA
Status: Suspended | Type: Observational
Why Stopped: The restrictions on research imposed for the COVID-19 pandemic prevented us from continuing recruitment and visits. At this stage our funding is not sufficient to continue enrollment so we will put the study in a hold pattern.
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 10-01329; 5R01HL080414-08 (NIH)
Record Dates: First submitted 2008-01-02; First posted 2008-01-16 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Sputum, whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Asthma: People who have been diagnosed with Asthma

SUMMARY:
The purpose of this study is to identify the causes of asthma that were not previously suspected, to better understand the effects of inhaled steroids on asthma and to identify new way to treat asthma.

DETAILED DESCRIPTION:
In this study, we will explore mechanisms of exacerbation in asthma by careful characterization studies in asthmatics presenting in acute severe exacerbation. Specifically, we will determine the frequency of secretor status in these subjects by blood and saliva testing, and we will also perform a detailed cellular and biochemical analysis of their airway secretions. We will collect airway secretions using two methods. One method will be to have subjects cough sputum into a clean plastic container. The other method only applies to asthmatics with near-fatal asthma requiring intubation and mechanical ventilation. In these asthmatics, we will collect airway secretions by tracheal aspirate using methods normally applied in their clinical care.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects with a history of asthma between the ages of 18 to 75 years.
2. Physician diagnosis of asthma.
3. Currently experiencing an acute exacerbation of asthma. This exacerbation may be severe necessitating treatment in the emergency room, ICU, or hospital ward.
4. Ability to provide informed consent.

Exclusion Criteria:

1. Lung disease other than asthma.
2. Females who are lactating or who are pregnant.
3. Use of recreational drugs in the 1 month preceding the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: emergency deparment, admitted patients in the ICU and inpatient wards
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2006-05 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
rheological measurements (viscosity and elasticity) in sputum from patients with acute severe asthma | 1-2 years

CONTACTS AND LOCATIONS:
Overall Officials: John V Fahy, M.D., M.Sc., Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Airway Clinical Research Center, San Francisco, California, United States

REFERENCES:
- See also: UCSF Airway Clinical Research Center website — http://acrc.ucsf.edu